CLINICAL TRIAL: NCT00585923
Title: A Multi-Center Clinical Investigation of Slotted Hole Versus Fixed Hole C-Tek™ Anterior Cervical Plates
Brief Title: Slotted Hole Versus Fixed Hole C-Tek
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of follow-up information
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS-014
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2010-03-26 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Herniated Disc; Radiculopathy; Spondylolysis
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy; Spondylolysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usage of Fixed hole C-Tek™ Plate (Active Comparator): Fixed Hole Plate - The fixed hole plate means that the screws do not move, restricting motion and providing additional stability
  Interventions: Device: Fixed hole C-Tek™ Plate
- Usage of Slotted hole C-Tek™ Plate (Active Comparator): Slotted Hole Plate - Bone screw translates while plate is stationary, which ultimately promotes grafts settling through load sharing.
  Interventions: Device: Slotted hole C-Tek™ Plate

INTERVENTIONS:
Device: Fixed hole C-Tek™ Plate — Fixed hole C-Tek™ Plate
  Arms: Usage of Fixed hole C-Tek™ Plate
Device: Slotted hole C-Tek™ Plate — Slotted hole C-Tek™ Plate
  Arms: Usage of Slotted hole C-Tek™ Plate

SUMMARY:
The purpose of this study is to compare the fusion rates between the EBI, LLC C-Tek™ Anterior Cervical Plate, Slotted Hole Design versus the Fixed Hole Design.

DETAILED DESCRIPTION:
This study's purpose is to compare the fusion rates between the EBI, LLC C-Tek™ Anterior Cervical Plate, Slotted Hole Design versus the Fixed Hole Design

ELIGIBILITY:
Inclusion Criteria:

1. Radiographic evidence of compressed cervical roots or cord by either ossified bony elements or herniated nucleus pulposus.
2. Symptomatic radiculopathy appropriate to compressed nerve root.
3. Cervical spondylosis as evidenced by reactive changes in the vertebral bodies about the interspace, and may be associated with chronic discopathy.
4. Primary anterior cervical spinal fusion (ACDF) performed using an anterior cervical plate and either a discectomy (Smith-Robinson technique) or a Corpectomy.
5. Adult male or female, 18 to 75 years of age.
6. The subject or his/her legal guardian is willing to consent to participate in this study.
7. The subject will be available for follow-up for a minimum of 24 months.

Exclusion Criteria:

1. Traumatic cervical injury.
2. Posterior augmentation or revision fusion.
3. Cervical fusion involving C1 and C2 vertebrae.
4. Cervical fusion involving more than three levels.
5. Previous spine surgery at the same levels as those that will be fixed with the C-Tek plate.
6. Systemic conditions: Spondylitis, Paget's disease, Rheumatoid arthritis, Infection within two weeks before surgery, Cancer, Renal disease or insufficiency with creatinine level above 2, Chronic use of steroids or other conditions that may affect bone metabolism
7. Subjects who are pregnant, nursing or plan to be pregnant within the next 24 months.
8. Mental or physical conditions that may preclude compliance with physician instruction or the study protocol.
9. Subjects who require non-steroidal medications chronically for other conditions.
10. Subject declines to cooperate with the follow-up schedule.
11. Subject or legal guardian refuses or is unable to sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2002-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Batts, Study Director — Biomet Spine
Locations (1):
- Spine Institute of Louisiana, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done through the population of Dr. Nunley's practice. Once Dr. Nunley decided that the patient was a candidate for cervical fusion, he discussed the study with the patient. After subject signed the informed consent subject was randomized to the Slotted Hole or the Fixed Hole C Tek™ Anterior Cervical Plate.
Pre-assignment Details: Patients were included in this study if the answer to all of the inclusion criteria was yes and the answer to all of the exclusion questions was no.
Groups:
- Fixed Hole C-Tek Plate: Fixed Hole C-Tek Plate for Anterior Cervical Discectomy & Fusion (ACDF)
- Slotted Hole C-Tek Plate: Slotted Hole C-Tek Plate for ACDF
Period: Overall Study
Arm/Group | Fixed Hole C-Tek Plate | Slotted Hole C-Tek Plate
Started | 56 | 59
Completed | 25 | 26
Not Completed | 31 | 33
Not completed — Physician decided not to continue | 31 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Hole C-Tek Plate | Slotted Hole C-Tek Plate | Total
Number analyzed (Participants) | 56 | 59 | 115
Age, Customized [Count of Participants; unit: Participants] — There were 5 patients in the fixed hole group and 2 patients in the slotted hole group who do not have calculated age due to missing information that we were unable to obtain from the clinical site
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 46 | 50 | 96
    >=65 years | 5 | 7 | 12
    Unknown | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.46 (10.26) | 50.03 (10.04) | 49.76 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 34 | 66
  Male | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Fusion Success
Description: The fusion criteria will include radiographic evidence of no motion at the affected levels on flexion/extension and evidence of bony bridging and no lucent lines on AP/lateral views.
  Fusion Grading
  "fused" "probably fused" "pseudarthrosis"
  This determination was made by Dr. Nunley and there was never any more specific details given on how the determination was made between fused and probably fused.
Time Frame: Last Follow-Up (Last follow-up ranged from no visit after surgery to 24 months of follow-up)
Population: Fusion Status is shown for the last office visit which the patient attended before the doctor withdrew from the study
Measure: Number; unit: participants
Arm/Group | Fixed Hole C-Tek Plate | Slotted Hole C-Tek Plate
Number analyzed (Participants) | 56 | 59
participants
  Solid Fused | 27 | 29
  Probably Fused | 15 | 22
  Pseudarthrosis (Failed Fusion) | 5 | 0
  No Fusion Result | 9 | 8

2. Secondary Outcome: Pain at Rest
Description: Pain is calculated by patient making an X on a visual analog scale (VAS) line at each visit. Mark on x is measured via a mm ruler. Number of Participants with the Level of Pain at Rest Improved, Maintained or Worsened from Baseline to "last follow-up visit". This is calculated by subtracting the pain at the last follow-up from the pain at the baseline visit. Best Case is 0 and worst case is 100.
Time Frame: Baseline and Last Follow-Up visit (Last follow-up ranged from no visit after surgery to 24 months of follow-up)
Measure: Number; unit: Participants
Arm/Group | Fixed Hole C-Tek Plate | Slotted Hole C-Tek Plate
Number analyzed (Participants) | 56 | 59
Participants
  Improved | 49 | 45
  Maintained | 1 | 2
  Worsened | 4 | 0
  No Pain Recorded at Last Visit | 2 | 12

3. Secondary Outcome: Pain With Activity
Description: Pain is calculated by patient making an X on a visual analog scale (VAS) line at each visit. Mark on x is measured via a mm ruler. Number of Participants with the Level of Pain with Activity Improved, Maintained or Worsened from Baseline to "last follow-up visit". This is calculated by subtracting the pain at the last follow-up from the pain at the baseline visit. Scores range from 0 to 100 with 0 being the best score.
Time Frame: Baseline and Last follow-up visit (Last follow-up ranged from no visit after surgery to 24 months of follow-up)
Measure: Number; unit: Participants
Arm/Group | Fixed Hole C-Tek Plate | Slotted Hole C-Tek Plate
Number analyzed (Participants) | 56 | 59
Participants
  Improved | 42 | 46
  Maintained | 1 | 1
  Worsened | 6 | 4
  No pain recorded at last visit | 7 | 8

4. Secondary Outcome: Neurological Status Change in Neurological Status Since Surgery.
Description: Patients were categorized as maintained, improved or decreased Neurological Status. This was assessed pre-operatively and at each follow-up visit but reported on last follow-up. Motor Function was measured at each cervical level Reflex Function (0: Not elicitable; 1: Elicited with reinforcement; 2: Normal; 3:Brisk; 4:Clonus, unsustained; 5: Clonus, sustained) was measured for Bicep, Brachioradialis, and Triceps Sensory Function (0: Sensation is absent; 1: Sensating is diminished; 2: Sensation is normal; 3: Sensation is present, but pathological, was measured at each cervical dermatome
Time Frame: Baseline and Last follow-up visit (Last follow-up ranged from no visit after surgery to 24 months of follow-up)
Measure: Number; unit: Participants
Arm/Group | Fixed Hole C-Tek Plate | Slotted Hole C-Tek Plate
Number analyzed (Participants) | 56 | 59
Participants
  Improved | 21 | 27
  Maintained | 17 | 16
  Decreased | 1 | 3
  Not Measured at last visit | 17 | 13

5. Secondary Outcome: Level of Function (Neck Disability Index)
Description: Number of patients who have an improved, maintained or decreased level of function based on the results of their NDI (Neck Disabillity Index) from surgery to last follow-up visit. The NDI scale ranges from 0-100. If a subject has a score of 0, it means that they have no limitations and no pain. This is calculated by subtracting the NDI at the last follow-up from the NDI at the baseline visit.
Time Frame: Baseline and Last follow-up visit (Last follow-up ranged from no visit after surgery to 24 months of follow-up)
Measure: Number; unit: Participants
Arm/Group | Fixed Hole C-Tek Plate | Slotted Hole C-Tek Plate
Number analyzed (Participants) | 56 | 59
Participants
  Improved | 39 | 43
  Maintained | 1 | 2
  Decreased | 8 | 7
  Not Measured at last visit | 8 | 7

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through the 24 mnth visit
Arm/Group | Fixed Hole C-Tek Plate | Slotted Hole C-Tek Plate
Serious Adverse Events (participants affected / at risk) | 2/56 | 0/59
Other Adverse Events (participants affected / at risk) | 1/56 | 0/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed Hole C-Tek Plate (N=56) | Slotted Hole C-Tek Plate (N=59)
Instrument Failure - Screw Breakage (Surgical and medical procedures) | 1 (1) | 0 (0) — Breakage of 2 screws
Instrument Failure - Screw Back-out (Surgical and medical procedures) | 1 (1) | 0 (0) — Screw backed out of the plate
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed Hole C-Tek Plate (N=56) | Slotted Hole C-Tek Plate (N=59)
Mild Wound Drainage (Infections and infestations) | 1 (1) | 0 (0) — Patient experienced a mild wound drainage

LIMITATIONS AND CAVEATS:
Early termination of this study because the doctor involved in the study decided that he did not want to participate in the study any more. The site also did not have very good follow-up on all of their patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No